CLINICAL TRIAL: NCT02541357
Title: Effects of Preoperative Relaxation and Intensified Surgery Education on Preoperative Wellbeing and Postoperative Complaints in Patients Undergoing Colorectal Surgery - a Randomized Controlled Trial
Brief Title: Preoperative Relaxation and Intensified Patient Surgery Education in Patients Undergoing Colorectal Surgery
Acronym: MBM_Colo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment insufficient
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Gustav Dobos, Principle Investigator, Universität Duisburg-Essen
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 15-6459 MBM Colorectal
Record Dates: First submitted 2015-09-01; First posted 2015-09-04 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Gastrointestinal Diseases
Keywords: Colorectal Surgery
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Usual care (No Intervention): Does not receive a specific study intervention
- preoperative relaxation program (Experimental): preoperative relaxation program
  Interventions: Behavioral: relaxation program
- preoperative surgery education (Experimental): single education unit to understand the complete surgical procedures
  Interventions: Behavioral: surgery education
- preop relaxation and surgery education (Experimental): preoperative relaxation program AND single education unit
  Interventions: Behavioral: relaxation program; Behavioral: surgery education

INTERVENTIONS:
Behavioral: relaxation program — relaxation and mindfulness techniques such as body scan, breathing meditation or imagination exercises
  1 week program, one introductory session and daily home practice
  Arms: preop relaxation and surgery education; preoperative relaxation program
Behavioral: surgery education — intensified education unit to reduce anxiety and stress, by using pictures and videos of rooms, and procedures of the planned surgery
  1 single unit in the week before the surgery
  Arms: preop relaxation and surgery education; preoperative surgery education

SUMMARY:
This study aims to test the effects of a Preoperative Relaxation intervention and an Intensified Surgery Patient Education on pre- and postoperative wellbeing and health in Patients Undergoing colorectal surgery.

DETAILED DESCRIPTION:
A former pilot study has shown that a preoperative relaxation program was effective in reducing preoperative anxiety. However the intervention was biased by concurrent pre-surgery education. Therefore this study aims to test the effects of a Preoperative Relaxation intervention and an Intensified Surgery Patient Education on pre- and postoperative wellbeing and health in Patients Undergoing colorectal surgery using a factorial design.

ELIGIBILITY:
Inclusion Criteria:

* referral for colorectal surgery
* preoperative anxiety at least 4/10 points on a numeric rating scale
* physical and mental capability to participant
* written informed consent

Exclusion Criteria:

* Emergency surgery
* known malignoma
* severe comorbidity
* severe psychological disorders
* immunosuppression
* coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
preoperative anxiety | day of surgery
  State Anxiety (STAI-S) (Spielberger 1970)
postoperative pain intensity | day after the surgery, before meditation
  numeric rating scale for pain at rest, pain at mobilization, coughing, washing, breathing and moving

SECONDARY OUTCOMES:
preoperative anxiety | day of surgery
  Trait Anxiety (STAI-T) (Spielberger 1970)
preoperative anxiety | day of surgery
  Amsterdam Preoperative Anxiety and Information Scale (APAIS) (Berth 2007)
preoperative anxiety | day of surgery
  Anaesthesia- and Surgery-dependent Preoperative Anxiety (ASPA) (Wetsch 2009)
postoperative disability | day after surgery
  interference of pain with movement, coughing, waking up at night and disturbed mood
postoperative disability | 2 days after surgery
  interference of pain with movement, coughing, waking up at night and disturbed mood
postoperative disability | 10 days after surgery
  interference of pain with movement, coughing, waking up at night and disturbed mood
postoperative fatigue | day after surgery
  Fatigue measured by 0-10 Numeric Rating Scale
postoperative fatigue | 2 days after surgery
  Fatigue measured by 0-10 Numeric Rating Scale
postoperative fatigue | 10 days after surgery
  Fatigue measured by 0-10 Numeric Rating Scale
postoperative nausea | Day after surgery
  Nausea measured by 0-10 Numeric Rating Scale
postoperative nausea | 2 days after surgery
  Nausea measured by 0-10 Numeric Rating Scale
postoperative nausea | 10 days after surgery
  Nausea measured by 0-10 Numeric Rating Scale
postoperative complications | 10 days after surgery
  Number of Participants With Treatment-Related Adverse Events
Satisfaction with care | 10 days after surgery
  Satisfaction with the operation, the hospital care on a visual analog scale each from 0 (not satisfied) to 100 (most satisfied)
Satisfaction with interventions | 10 days after surgery
  Satisfaction with interventions on a visual analog scale each from 0 (not satisfied) to 100 (most satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof, MD, Principal Investigator — Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, University of Duisburg-Essen
Locations (1):
- Abteilung für Allgemein-, Viszeral-, Gefäßchirurgie und Koloproktologie, Johanniter-Krankenhaus Rheinhausen, Duisburg, Germany

IPD SHARING:
Plan to Share IPD: No
Study has been terminated